CLINICAL TRIAL: NCT04901962
Title: Prospective Multicentre Study to Evaluate the Clinical Performance and Safety of Innovative, Made-to-measure Compression Garments in Daily Routine
Brief Title: Study to Evaluate Made-to-measure Compression Garments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BSN Medical GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C2612
Record Dates: First submitted 2021-05-17; First posted 2021-05-26 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2022-02

CONDITIONS: Lymphedema
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JOBST® Confidence compression garments (Experimental): The CE-marked class I medical devices JOBST® Confidence compression garments for lower and upper extremities will be tested under routine conditions according to their selected intended use. Subjects will be treated with either thigh-high compression stockings (AG) or arm compression garments without hand part (CG1), depending on their indication.
  Interventions: Device: JOBST® Confidence compression garments

INTERVENTIONS:
Device: JOBST® Confidence compression garments — JOBST® Confidence (JC) compression garments will be used for daytime treatment of leg or arm lymphedema. JC compression garments exert a specific therapeutic external, physical compression level and are therefore intended to use for the management of edema. JC comprise non-invasive medical devices with no direct contact with injured skin or mucous membranes and are intended for use on intact skin only.

SUMMARY:
The primary objective is to collect real-life data to evaluate the clinical performance and safety of innovative, made-to-measure, flat knitted, CE-marked compression garments for daytime treatment of leg or arm lymphedema (ISL stage I-II) in daily routine by analysing performance parameters and safety parameters reported during the investigation.

DETAILED DESCRIPTION:
The secondary objective is to evaluate (1) patients' quality of life QoL before and after having tested JOBST Confidence and (2) patient satisfaction focussing on patient reported outcomes of previously worn garments and JOBST® Confidence by analysing patient questionnaires parameters completed at the beginning and in the end of the wearing period.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form
2. Men, women or diverse aged 18 years or up to 70 years with full legal competence
3. Patient is mentally and physically able to participate in the study
4. Capability to understand the subject information and to provide conscious informed consent
5. Capability and willingness to follow protocol requirements
6. All female or diverse subjects of childbearing potential must agree to use a reliable method of contraception with a Pearl-Index of less than 1% per year when used consistently and correctly* (*such as hormone implants,injectables, combined oral contraceptives (combined gestagen-estrogen pills), some intra uterine devices (IUDs), surgically sterility (hysterectomy or tubal ligation), sexual abstinence or vasectomized partner for at least 4 weeks)
7. Mild to moderate lymphedema of the lower and/or upper extremities (ISL stage I or II)
8. Indication and possibility of treatment with a flat-knitted compression garment during the day
9. Patients who are familiar with wearing compression garments
10. Indicated Complete Decongestive Therapy Phase II (Maintenance phase)
11. Willingness to wear the study product at least 5 days a week for at least 6 hours a day

Exclusion Criteria:

1. Pregnant or lactating women or diverse subjects
2. Alcohol abuse (mentioned by the patient and/or suspected by the investigator)
3. Drug abuse (mentioned by the patient and/or suspected by the investigator)
4. Patients who need a different compression class (higher or lower than CCL 2)
5. Pronounced skin folds
6. Pronounced shape distortions
7. cG (lymphatic measure of the thigh) >90 cm for AG stocking
8. Indicated Complete Decongestive Therapy Phase I
9. Known allergy or intolerance to one or more components of the product
10. Advanced arterial insufficiency including ischemia
11. Uncontrolled congestive heart failure
12. Untreated septic phlebitis
13. Phlegmasia coerulea dolens
14. Immobility (confinement to bed).
15. Conditions in which increased venous and lymphatic return is not desired.
16. Weeping dermatosis
17. Cutaneous infections
18. Severely compromised skin sensibility and impaired sensitivity of the limb
19. Advanced peripheral neuropathy
20. Rheumatoid arthritis
21. Complex regional pain syndrome (CRPS, M. Sudeck)
22. Malignant lymphedema
23. Gangrene
24. Sponsors or manufacturers staff
25. Open wounds in the test area
26. Diuretics, except low doses for treatment of hypertension (≤ 12.5 mg Hydrochlorothiazide)
27. Nephrotic syndrome

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2021-07-21 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
Clinical performance: circumference of the edema | change from baseline after a treatment duration of 7, 14, and 21 days
  Circumference measurements at selected points of the limb (taken manually using measuring tape) [cm]
Clinical performance: edema status | change from baseline after a treatment duration of 7, 14, and 21 days
  Evaluation of edema (visual inspection and palpitation) according to standardized criteria

SECONDARY OUTCOMES:
Quality of Life assessed by patient questionnaire | assessed before treatment and after 21 days of treatments with JC
  extend of restrictions regarding work due to the lymphoedema (indicated on a 5-point scale)
Quality of Life assessed by patient questionnaire | assessed before treatment and after 21 days of treatments with JC
  extend of restrictions regarding leisure time due to the lymphoedema (indicated on a 5-point scale)
Quality of Life assessed by patient questionnaire | assessed before treatment and after 21 days of treatments with JC
  extend of restrictions regarding psychological well-being due to the lymphoedema (indicated on a 5-point scale)
Patient satisfaction assessed by patient questionnaire | assessed before treatment and after 21 days of treatments with JC
  Comparison of patient reported outcomes regarding previously worn compressions garments and JC

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Hirsch, Dr. med., Principal Investigator — Praxis für Innere Medizin und Gefäßkrankheiten
Locations (4):
- Germany (4):
  - Gefäßkrankheiten Rhein-Ruhr, Essen, North Rhine-Westphalia
  - Dr. Hans-Walter Fiedler, Werl, North Rhine-Westphalia
  - Praxis für Innere Medizin und Gefäßkrankheiten, Halle, Saxony-Anhalt
  - Dr. med. Jörg Schleinitz Facharzt für Allgemeinmedizin, Lützen, Saxony-Anhalt

IPD SHARING:
Plan to Share IPD: No